CLINICAL TRIAL: NCT01881581
Title: A Phase I Double-Blind Study to Evaluate the Safety and Immunogenicity of HIV Prime/Boost Vaccine Using DNA and MVA for HIV-1/AIDS
Brief Title: Safety and Immunogenicity of Recombinant HIV Vaccines for HIV/AIDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Beijing Ditan Hospital (Other); National Institutes for Food and Drug Control, China (Other)
Responsible Party: Principal Investigator, Yi Zeng, Departement Director, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDCPChina001
Record Dates: First submitted 2013-06-16; First posted 2013-06-19 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Therapeutic; Vaccine; HIV; MVA; DNA
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Lower dose DNA or Placebo (Experimental): 2.0 mL lower dose D-GPEi (0.5mg) or Saline solution at weeks 0
  Interventions: Biological: Saline Solution; Biological: D-GPEi
- Medium dose DNA or Placebo (Experimental): 2.0 mL medium dose D-GPEi (2mg) or Saline solution at weeks 0
  Interventions: Biological: Saline Solution; Biological: D-GPEi
- High dose DNA or Placebo (Experimental): 2.0 mL high dose D-GPEi (4mg) or Saline solution at weeks 0
  Interventions: Biological: Saline Solution; Biological: D-GPEi
- Lower dose MVA or Placebo (Experimental): 100μL lower dose M-GPE (3×10^7pfu) or Saline solution at weeks 0
  Interventions: Biological: Saline Solution; Biological: M-GPE
- Medium dose MVA or Placebo (Experimental): 100μL medium dose M-GPE (1×10^8pfu) or Saline solution at weeks 0
  Interventions: Biological: Saline Solution; Biological: M-GPE
- High dose MVA or Placebo (Experimental): 300μL high dose M-GPE (3×10^8pfu) or Saline solution at weeks 0
  Interventions: Biological: Saline Solution; Biological: M-GPE
- Low dose DNA+MVA or Placebo control (Experimental): The dose below the maximum tolerated dose of D-GPEi or 2.0 mL Saline solution at week 0,1; The dose below the maximum tolerated dose of M-GPE or 100/300μL Saline solution at week 2,3
  Interventions: Biological: Saline Solution; Biological: D-GPEi; Biological: M-GPE
- High dose DNA+MVA or Placebo control (Experimental): The maximum tolerated dose of D-GPEi or 2.0 mL Saline solution at week 0,1;The maximum tolerated dose of M-GPE or 100/300μL Saline solution at week 2,3
  Interventions: Biological: Saline Solution; Biological: D-GPEi; Biological: M-GPE

INTERVENTIONS:
Biological: Saline Solution — Saline Solution is used as control in all arms.
Biological: D-GPEi — D-GPEi is used in Arm A,B,C,G and H.
  Arms: High dose DNA or Placebo; High dose DNA+MVA or Placebo control; Low dose DNA+MVA or Placebo control; Lower dose DNA or Placebo; Medium dose DNA or Placebo
Biological: M-GPE — M-GPE is used in Arm D,E,F,G and H
  Arms: High dose DNA+MVA or Placebo control; High dose MVA or Placebo; Low dose DNA+MVA or Placebo control; Lower dose MVA or Placebo; Medium dose MVA or Placebo

SUMMARY:
This is a randomized, double-blind placebo-controlled dose-escalation clinical trial to evaluate the safety and the immunogenicity of DNA and modified vaccinia virus Ankara (MVA) HIV-1 vaccines in subjects receiving stable highly active antiretroviral therapy (HAART) who have an HIV-1 RNA < 50 copies/mm3 and CD4+ T cells count ≥ 350 cells/mm3.

DETAILED DESCRIPTION:
HIV-infected patients treated with antiretroviral therapy for prolonged periods of time may show decreased levels of HIV-specific immune responses. In these patients, a prime-boost vaccine strategy may induce both humoral and cell-mediated immunity. The hypothesis of this study is that the vaccine strategy selected will be both safe and immunogenic in the patient population being tested.

Patients continue antiretroviral medications throughout the course of this study. Three groups of patients receive dose-escalation (0.5mg, 2mg or 4mg) intramuscular injections of DNA vaccine (D-GPEi) respectively, the other three groups of patients receive dose-escalation (3×10^7pfu, 1×10^8pfu or 3×10^8pfu) intradermal injections of MVA vaccine (M-GPE), two weeks post immunization of lower dose, if the vaccine is safe and well tolerant, the next dose of immunization will begin. After the maximum tolerated dose of DNA and MVA is identified, DNA prime/ MVA boosting will be tested in another two groups of patients. Lower or the maximum tolerated dose of D-GPEi was used at week 0 and 1, lower or the maximum tolerated dose of M-GPE was used at week 2 and 3, patients are monitored for safety 72 hours after each immunization. In addition, each patient records adverse events in a diary. Patients have regular physical exams, pregnancy tests, and blood drawn for virologic and immunologic assessments. The induction of HIV-specific responses will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Are willing to participate this study and available for follow-up for the duration of the study.
* Men and women aged 18-50 years.
* Are HIV-positive.
* Have been taking stable anti-HIV drugs for at least 6 months.
* CD4 count ≥ 350 cells/mm3
* Plasma viral load < 50 copies/ml.
* Willing to use acceptable forms of contraception at least 21 days prior to first vaccination until 56 days after the last vaccination.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* History of previous vaccination with an HIV-1 vaccine.
* Use of immunoinhibitory agents, such as corticosteroids or cytotoxic drugs by oral administration, injection route or inhalation route within 6 months of study entry (But corticosteroids used for allergic rhinitis and skin topical application of corticosteroids were not included); Use of immunomodulatory agents including but not limited to interleukin-2(IL-2） and granulocyte-macrophage colony-stimulating factor (GM-CSF) within 30 days of study entry.
* Use of blood products within 3 months of study entry.
* Use of other experimental drugs within 3 months of study entry.
* Any immunization within 3 months of study entry.
* Comply with any of the following items： Active pulmonary tuberculosis； History of serious adverse reaction to other vaccines； Serious asthma； Have untreated thyroid disease; Syphilis
* Laboratory values（Comply with any of the following items）:

Hemoglobin < 100 g/L (male subjects)，<90 g/L (female subjects)； Absolute neutrophil count ≤ 1000 cells/mm3； Serum creatinine ≥15 mg/L，endogenous creatinine clearance rate <50 ml/min； alanine aminotransferase（ALT）, aspartate aminotransferase(AST) ≥3× upper limit of normal range； Total bilirubin ≥2× upper limit of normal range

* Clinically significant electrocardiogram changes.
* Hypertension ( If it is well controlled by medication and is less than 150/100mmHg , should not be excluded) and other cardiac disease；
* Any medical, psychiatric, social condition, occupational reason judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of local and systemic adverse events | 8 months
  To evaluate the safety and tolerance of a DNA and a replication-defective MVA vaccine expressing HIV-1 gag-pol and env in HIV-1 infected subjects on highly active antiretroviral therapy.
  Frequency and severity of adverse events, laboratory abnormalities, and local and systemic reactogenicity signs and symptoms following vaccinations

SECONDARY OUTCOMES:
Immunogenicity of vaccine | 14 months
  Changes in CD4+ and CD8+ T-cell counts pre- and post-immunization and between the vaccine and placebo groups Changes in viral load pre- and post-immunization and between the vaccine and placebo groups Magnitude and breadth of HIV-1 specific CD8+ T cell responses as determined by interferon-γ(IFN-γ) enzyme-linked immunospot (ELISPOT) using overlapping HIV peptides for gag, pol and env Changes in HIV-1 Gp160-specific antibody responses pre- and post-immunization and between the vaccine and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Xingwang Li, M.D., Principal Investigator — Beijng Ditan Hospital of Capital Medical University; Rongmeng Jiang, M.D., Principal Investigator — Beijng Ditan Hospital of Capital Medical University; Yi Zeng, Principal Investigator — National Institute for Viral Disease Control and Prevention, China CDC; Xia Feng, Ph.D, Principal Investigator — National Institute for Viral Disease Control and Prevention, China CDC; Ke Xu, Ph.D, Principal Investigator — National Institute for Viral Disease Control and Prevention, China CDC
Locations (1):
- Beijing Ditan Hospital of Capital Medical University, Beijing, China